CLINICAL TRIAL: NCT02673099
Title: The Benefit of Оn-Line High Convection Volume Hemodiafiltration Treatment Versus High Flow Dialysis on Reduction of Oxidative Stress and Health Related Quality of Life in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0082-13
Record Dates: First submitted 2016-01-30; First posted 2016-02-03 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: End Stage Renal Disease
Keywords: HDF online; ESRD; Hemodialysis; oxidative stress; quality of life; Hemodialysis treatment
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HDF online (Other): All patients were started on HF (high-flux) hemodialysis. After 6 months they were then treated by HDF online.
  Interventions: Procedure: HDF online

INTERVENTIONS:
Procedure: HDF online — Hemodialysis by the HDF online method

SUMMARY:
Introduction: Patients with end stage renal disease are exposed to metabolic and hemodynamic complications due to the disease itself and as a result of the dialysis treatment related complications. Uremic toxins due to their middle molecular weight are not effectively removed during Hemodialysis. Their accumulation leads to chronic oxidative stress and chronic inflammation state associated with increased morbidity and mortality. In addition, during each dialysis session oxidative stress (OS) and inflammation are provoked once blood interacts with the dialyzer.

In recent years the use of Online Hemodiafiltration (OL- HDF) has entered in order to enable better uremic toxins clearance. This a relatively new method of therapy that allows a larger volume of blood filtration during a single dialysis therapy compared with standard hemodialysis. It combines diffusion with convection to clear middle molecular weight substances more effectively compared with Hemodialysis. This method was found to reduce rates of cardiovascular morbidity and mortality among dialysis patients.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether dialysis by high convection volume OL HDF reduces oxidative stress and inflammation levels, improving hemodynamic stability and metabolic complications compared to dialysis with High Flux (HF) membranes.

Methods: After a rush in period of 3 month with HF membranes, 45 dialysis patients were treated with HF for 6 months and then converted to 6 months of OL HDF treatment. The hemodynamic stability was measured during treatment throughout all the study and Quality of life was assessed by a reliable and valid tool developed and adapted specifically for ESRD population according to Kidney Disease Quality of Life Short Form (KDQOL- SF).

We propose to measure biomarkers of inflammation and oxidative stress in all blood samples collected at the end of each period for the following ( The number of blood samples to be analyzed: 45 patients 3 samples per patient total of 135 samples ).

* Total glycated proteins in relation to total proteins and to oncotic pressure of the samples. We have shown that the oncotic pressure can serve as a better measure of albumin concentrations than the albumin measured in routine clinical laboratories3.
* Albumin detection index4 and levels of albumin, as a measure of oxidation and inflammation (negative acute phase protein).
* Levels of Beta2m.
* Levels of Klotho: It was shown that reduced serum soluble Klotho is associated with all-cause mortality, even after adjusting for confounding variables, implying that the level of serum soluble Klotho plays a role as a predictive indicator of overall mortality in patients with ESRD.
* Levels of myeloperoxidase (MPO), a products of neutrophils degranulation due to activation by the dialysis treatment.
* Oxidation reduction potential (ORP), a global measure of all oxidant and antioxidant activity (A new instrument introduced in our research laboratory)
* Advanced oxidation protein products (AOPP) , a measure of total protein oxidation

Implication: The study will examine whether OL-HDF dialysis with high convection volume is associated with a reduction of oxidative stress and inflammation markers and improvement in the quality of life of dialysis patients. The results of this study will encourage the use of this new treatment mode in order to reduce the high morbidity resulting from OS and inflammation among these patients.

ELIGIBILITY:
Inclusion Criteria:

* On chronic hemodialysis more than 3 months

Exclusion Criteria:

* No exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Improvement of quality of life | 1 year

SECONDARY OUTCOMES:
Oxidative stress reduction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No